CLINICAL TRIAL: NCT02407626
Title: Optimierung Der Kardioprotektion Durch Inhalative Anästhetika Eine Untersuchung Bei Patienten Mit Diabetes Mellitus während Off-pump Herzchirurgie
Brief Title: Optimization of Cardioprotection in Diabetic Patients Undergoing Cardiac Surgery
Acronym: OPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very low patient recruitment, changed insurance requirements
Sponsor: Triemli Hospital (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Christoph K Hofer, Prof. Dr. med., Triemli Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STZ-IFA-0115
Record Dates: First submitted 2015-03-18; First posted 2015-04-03 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Ischemia
Keywords: ischemia; cardiac surgery; volatile anesthetic; total intravenous anesthesia
MeSH Terms: conditions — Myocardial Ischemia; Ischemia | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Volatile anesthesia for elective cardiac surgery
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): Total intravenous anesthesia for elective cardiac surgery
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Total intravenous anesthesia is a clinical standard procedure
  Arms: Propofol
Drug: Sevoflurane — Volatile anesthesia is a clinical standard procedure
  Arms: Sevoflurane

SUMMARY:
This study evaluates the myocardial protection against perioperative ischemia comparing two standard anesthetic regimes in diabetic patients undergoing elective cardiac surgery. Half of the patients will receive volatile anesthesia while the other half will receive total intravenous anesthesia. Primary and secondary outcome parameters will be assessed after induction of anesthesia, at the end of the procedure and postoperative day 1 to 3.

DETAILED DESCRIPTION:
Volatile anaesthetics such as Sevoflurane have shown to have a protective effect regarding myocardial ischemia in the perioperative setting - the so-called "preconditioning". However the observed response of preconditioning in clinical trials is not consistent.

An increased perioperative insulin resistance especially in diabetic patients resulting in an increased postoperative morbidity and mortality may be responsible for these findings.

In an animal model, the use of propofol that is being routinely applied for general anesthesia was associated with a change of the insulin receptor substrate via phosphorylation and thus a change of insulin resistance.

Avoiding a total intravenous anesthesia and applying a volatile anesthesia may result in an increased cardioprotective effect by a reduction of the perioperative insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Elective cardiac surgery

Exclusion Criteria:

* Emergency procedures
* Preop myocardial infarction
* Preop cardiac failure
* Preop renal replacement therapy

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Biomarker NT-proBNP | 1. after induction of anesthesia 2. after chest closure 3.-5. postoperative day 1, day 2, day 3
  Difference between volatile anesthesia and total intravenous anesthesia

SECONDARY OUTCOMES:
Receptor Substrate phosphorylization (IRS-1)/PP2A | 1. beginning of cardiac surgery, 2. end of cardiac surgery
  Difference between volatile anesthesia and total intravenous anesthesia
Expression of TNF/IL1beta and microRNA (miR144, miR125b, miR208a) | 1. beginning of cardiac surgery, 2. end of cardiac surgery
  Difference between volatile anesthesia and total intravenous anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zollinger, MD, Study Chair — Institute of Anesthesiology and Intensive Care Medicine Triemli City Hospital Zurich
Locations (1):
- Triemli City Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Julier K, da Silva R, Garcia C, Bestmann L, Frascarolo P, Zollinger A, Chassot PG, Schmid ER, Turina MI, von Segesser LK, Pasch T, Spahn DR, Zaugg M. Preconditioning by sevoflurane decreases biochemical markers for myocardial and renal dysfunction in coronary artery bypass graft surgery: a double-blinded, placebo-controlled, multicenter study. Anesthesiology. 2003 Jun;98(6):1315-27. doi: 10.1097/00000542-200306000-00004. PMID 12766638
- [Background] Lucchinetti E, Hofer C, Bestmann L, Hersberger M, Feng J, Zhu M, Furrer L, Schaub MC, Tavakoli R, Genoni M, Zollinger A, Zaugg M. Gene regulatory control of myocardial energy metabolism predicts postoperative cardiac function in patients undergoing off-pump coronary artery bypass graft surgery: inhalational versus intravenous anesthetics. Anesthesiology. 2007 Mar;106(3):444-57. doi: 10.1097/00000542-200703000-00008. PMID 17325502
- [Background] Piriou V, Mantz J, Goldfarb G, Kitakaze M, Chiari P, Paquin S, Cornu C, Lecharny JB, Aussage P, Vicaut E, Pons A, Lehot JJ. Sevoflurane preconditioning at 1 MAC only provides limited protection in patients undergoing coronary artery bypass surgery: a randomized bi-centre trial. Br J Anaesth. 2007 Nov;99(5):624-31. doi: 10.1093/bja/aem264. Epub 2007 Oct 3. PMID 17913754
- [Background] Zaugg M, Lucchinetti E, Uecker M, Pasch T, Schaub MC. Anaesthetics and cardiac preconditioning. Part I. Signalling and cytoprotective mechanisms. Br J Anaesth. 2003 Oct;91(4):551-65. doi: 10.1093/bja/aeg205. PMID 14504159
- [Background] Zaugg M, Lucchinetti E, Garcia C, Pasch T, Spahn DR, Schaub MC. Anaesthetics and cardiac preconditioning. Part II. Clinical implications. Br J Anaesth. 2003 Oct;91(4):566-76. doi: 10.1093/bja/aeg206. PMID 14504160
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Lou PH, Lucchinetti E, Zhang L, Affolter A, Gandhi M, Zhakupova A, Hersberger M, Hornemann T, Clanachan AS, Zaugg M. Propofol (Diprivan(R)) and Intralipid(R) exacerbate insulin resistance in type-2 diabetic hearts by impairing GLUT4 trafficking. Anesth Analg. 2015 Feb;120(2):329-40. doi: 10.1213/ANE.0000000000000558. PMID 25437926
- [Background] Whittington RA, Virag L, Marcouiller F, Papon MA, El Khoury NB, Julien C, Morin F, Emala CW, Planel E. Propofol directly increases tau phosphorylation. PLoS One. 2011 Jan 31;6(1):e16648. doi: 10.1371/journal.pone.0016648. PMID 21304998
- [Background] Swart MJ, De Jager WH, Kemp JT, Nel PJ, Van Staden SL, Joubert G. The effect of the metabolic syndrome on the risk and outcome of coronary artery bypass graft surgery. Cardiovasc J Afr. 2012 Aug;23(7):400-4. doi: 10.5830/CVJA-2012-055. PMID 22914999
- [Background] Wang L, Ko KW, Lucchinetti E, Zhang L, Troxler H, Hersberger M, Omar MA, Posse de Chaves EI, Lopaschuk GD, Clanachan AS, Zaugg M. Metabolic profiling of hearts exposed to sevoflurane and propofol reveals distinct regulation of fatty acid and glucose oxidation: CD36 and pyruvate dehydrogenase as key regulators in anesthetic-induced fuel shift. Anesthesiology. 2010 Sep;113(3):541-51. doi: 10.1097/ALN.0b013e3181e2c1a1. PMID 20683255